CLINICAL TRIAL: NCT01575106
Title: A Brain Imaging Study of the Analgesic Effect of Lidocaine and the Hyperalgesic Effect of Capsaicin
Brief Title: The Neurobiology of Expectancy and Pain Perception
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Jian Kong, Assistant Professor, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2011P000663
Record Dates: First submitted 2012-02-24; First posted 2012-04-11 (Estimated); Results first posted 2017-10-13 (Actual); Last update posted 2017-10-13 (Actual); Status verified 2017-01

CONDITIONS: Pain
MeSH Terms: conditions — Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Arm 1 (Experimental): There is only one cohort in this study. All subjects receive the same intervention, the application of heat pain using TSA or CHEPS.
  Interventions: Device: Heat pain applied using TSA or CHEPS

INTERVENTIONS:
Device: Heat pain applied using TSA or CHEPS — TSA-2001 Thermal Sensory Analyzer (Medoc LTD Advanced Medical Systems) or the Pathway Medoc (CHEPS model, Contact Heat-Evoked Potential Stimulator, Medoc LTD Advanced Medical Systems)

SUMMARY:
This study will use using fMRI (functional Magnetic Resonance Imaging) to elucidate how contextual learning/expectation relieves or aggravates pain experience in the same cohort of subjects and the same study session.

ELIGIBILITY:
Inclusion Criteria:

* a) Healthy male and female adults aged 21-50
* b) No contraindications to fMRI scanning
* c) Right handed

Exclusion Criteria:

* a) Current or past history of major medical, neurological, or psychiatric illness
* b) Pregnancy or breast feeding, menopause, and irregular menstrual cycles (length of cycle must be within 26 to 32 days)
* c) Claustrophobia
* d) History of head trauma
* e) History of impaired elimination
* f) Instability of responses to experimental pain (see Study Procedures Section)
* g) Use of psychotropic drugs, hormone treatments (including hormonal birth control) within 1 year
* h) Non-fluent speaker of English

Ages: 21 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 38 (Actual)
Dates: Start 2012-06; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jian Kong, MD,eq/MS/MPH, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Charlestown, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Heat Pain: There is only one cohort in this study. All subjects receive the same intervention, the application of heat pain using TSA or CHEPS.
  Heat pain applied using TSA or CHEPS: TSA-2001 Thermal Sensory Analyzer (Medoc LTD Advanced Medical Systems) or the Pathway Medoc (CHEPS model, Contact Heat-Evoked Potential Stimulator, Medoc LTD Advanced Medical Systems)
Period: Overall Study
Arm/Group | Heat Pain
Started | 38
Completed | 24
Not Completed | 14

BASELINE CHARACTERISTICS:
Arm/Group | Heat Pain
Number analyzed (Participants) | 24
Age, Continuous [Mean (Standard Deviation); unit: years] | 26.5 (6.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 13

OUTCOME MEASURES:

1. Primary Outcome: Subjective Response to Pain (0-20 Visual Analogue Scale)
Description: Subjects received heat pain before and after the application of a neutral cream (told one application of neutral cream was lidocaine, one was capsaicin, and one was neutral) and rated pain intensity on a 0-20 Visual Analogue Scale (0-no pain, 20-intolerable pain). We only measure this outcome measure in session 3. The pain intensity for each cream was averaged amongst all participants for both the pre and post treatment in session 3. Subjects have up to 3 weeks to complete the 3 sessions.
Time Frame: Weeks 1-3
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Heat Pain
Number analyzed (Participants) | 24
units on a scale
  Pre-treatment placebo Lidocaine | 10.7 (2.4)
  Pre-treatment placebo capsaicin | 11 (1.8)
  Pre-treatment neutral | 11.2 (2.0)
  Post-treatment placebo lidocaine | 8.1 (3)
  Post-treatment placebo capsaicin | 12.2 (2.6)
  Post-treatment neutral | 10.8 (2.3)

2. Primary Outcome: fMRI Signal Changes in the Dorsal Anterior Cingulate Cortex
Description: We used fMRI to investigate the signal changes associated with administration of identical pain stimuli before (pre) and after the treatment (post) with different creams in session 3. It is important to note that the subjects had multiple weeks to complete the study, but this measure was only taken during one session. The change was calculated from two time points as the value at the later time point (post treatment) minus the value at the earlier time point (pre treatment).
Time Frame: Week 4
Population: The neutral cream is omitted from the data table below because we were only concerned about the direct comparison between positive expectancy ("Lidocaine") and negative expectancy ("Capsaicin") conditions. Data were only collected for the Lidocaine and Capsaicin creams.
Measure: Mean (Standard Deviation); unit: Post-Pre treatment peak beta
Arm/Group | Heat Pain
Number analyzed (Participants) | 24
Post-Pre treatment peak beta
  Lidocaine | 0.2 (0.18)
  Capsaicin | 0.3 (0.3)

ADVERSE EVENTS:
Groups:
- Heat Pain: All subjects receive the same intervention, the application of heat pain using TSA or CHEPS.
  Heat pain applied using TSA or CHEPS: TSA-2001 Thermal Sensory Analyzer (Medoc LTD Advanced Medical Systems) or the Pathway Medoc (CHEPS model, Contact Heat-Evoked Potential Stimulator, Medoc LTD Advanced Medical Systems)
- Cream: All subjects were told they would receive lidocaine, capsaicin, and neutral cream on their forearm, but in reality they only received neutral cream (regular moisturizing lotion).
Arm/Group | Heat Pain | Cream
All-Cause Mortality (participants affected / at risk) | 0/38 | 0/38
Serious Adverse Events (participants affected / at risk) | 0/38 | 0/38
Other Adverse Events (participants affected / at risk) | 1/38 | 0/38
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Heat Pain (N=38) | Cream (N=38)
Skin and tissue disorders (Skin and subcutaneous tissue disorders) | 1 | 0 — itching, tenderness, and burning

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No